CLINICAL TRIAL: NCT04788095
Title: Assessing Feasibility of an App-Based Mindfulness Intervention for Patients With Metastatic Renal Cell Carcinoma
Brief Title: App-Based Mindfulness Intervention for the Improvement of Quality of Life in Patients With Metastatic Renal Cell Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20310; NCI-2020-10496 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20310 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-12-01; First posted 2021-03-09 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Renal Cell Carcinoma; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device feasibility (app-based mindfulness program) (Experimental): Patients participate in a mindfulness-based program by using the Am app for 20-30 minutes every day, a minimum of 4 days each week over 4 weeks.
  Interventions: Behavioral: Behavioral Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Participate in an app-based mindfulness program
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial tests the feasibility of an application (app)-based mindfulness intervention and its effect on improving quality of life in patients with renal cell cancer that has spread to other places in the body (metastatic). This trial aims to see whether an app-based mindfulness intervention may help patients cope with their disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess feasibility of the Am mindfulness app in metastatic renal cell carcinoma (mRCC) patients, with respect to accrual, adherence and engagement in program.

II. To assess preliminary effects of app-based mindfulness intervention in patients with metastatic renal cell carcinoma (mRCC) (the Am Mindfulness-Based Cancer Survivorship [MBCS] Journey), on psychosocial outcomes (e.g., anxiety, distress, fear of cancer recurrence), as well as overall quality of life (QOL) and fatigue, among patients with mRCC.

OUTLINE:

Patients participate in a mindfulness-based program by using the Am app for 20-30 minutes every day, a minimum of 4 days each week over 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Sufficiently fluent in English
* Cytologically or pathologically verified diagnosis of renal cell carcinoma (RCC)
* Evidence of metastatic disease (including at a minimum computed tomography [CT] of the chest, abdomen and pelvis for staging)
* Undergoing immunotherapy
* A "moderate" or greater fear of cancer progression, as demonstrated by an Fear of Cancer Recurrence-7 (FCR-7) score of >= 17
* A fear of cancer progression, as demonstrated by a Patient Reported Outcomes Measurement Information System (PROMIS)-Anxiety score >= 13
* Have smart phone with internet access
* Not suffering from current major depressive disorder, bipolar disorder or other psychiatric disorder
* Not currently engaging in meditation one or more times per week within the previous year
* Has not participated in an mindfulness-based cancer recovery (MBCR) or mindfulness-based stress reduction (MBSR) program in the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility metric 1 | 3 months
  At least 90% of desired accrual is reached within 3 months (Yes or No)
Feasibility metric 2 | 3 months
  At least 70% of patients are able to complete at least 2 of 4 intended intervention sessions for at least 2 of 4 weeks (Yes or No)
Feasibility metric 3 | 3 months
  At least 70% of patients have at least 2 of 4 evaluable time points for the 4 assessments for Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety and Fear of Cancer Recurrence. (Yes or No)
Feasibility metric 4 | 3 months
  At least 70% of patients have at least 2 of 4 evaluable time points for the 4 assessments for Patient Reported Outcomes Measurement Information System (PROMIS) depression. (Yes or No)
Fear of Cancer Recurrence-7 | 3 months
  7-item scale that assesses the degree of FCR, with a cutoff score of 17 or above indicative of moderate and a cutoff score of 27 or above indicative of severe FCR. Reported as low, moderate, severe. Count and percentages provided for each level.
PROMIS Emotional Distress: Anxiety | 3 months
  This 8-item measure assesses symptoms of anxiety on a 5-point scale (1=never, 5=always). Scores range from 7-35 with higher scores indicating greater severity of anxiety. Data reported as continuous measure: means, standard deviation/ median range to be provided.
PROMIS Emotional Distress: Depression | 3 months
  This 8-item measure assesses symptoms of depression on a 5-point scale (1=never, 5=always). Scores range from 8-40 with higher scores indicating greater severity of depression. Data reported as continuous measure: means, standard deviation/ median range to be provided.
Functional Assessment of Chronic Illness Therapy-General (FACT-G): Overall | 3 months
  A 27-item self-related scale measure QoL across four domains of 'well-being' (physical, social/family, emotional and functional) on a 4-point Likert scale. Scores range from 0-108 for the total score. Data reported as continuous measure: means, standard deviation/ median range to be provided.
Functional Assessment of Chronic Illness Therapy-General (FACT-G): Physical | 3 months
  A 27-item self-related scale measure QoL across four domains of 'well-being' (physical, social/family, emotional and functional) on a 4-point Likert scale. Scores range from 0-28 for the physical. Data reported as continuous measure: means, standard deviation/ median range to be provided.
Functional Assessment of Chronic Illness Therapy-General (FACT-G): Social/ Family | 3 months
  A 27-item self-related scale measure QoL across four domains of 'well-being' (physical, social/family, emotional and functional) on a 4-point Likert scale. Scores range from 0-28 for the social/family. Data reported as continuous measure: means, standard deviation/ median range to be provided.
Functional Assessment of Chronic Illness Therapy-General (FACT-G): Functional | 3 months
  A 27-item self-related scale measure QoL across four domains of 'well-being' (physical, social/family, emotional and functional) on a 4-point Likert scale. Scores range from 0 to 28 for the functional subscales. Data reported as continuous measure: means, standard deviation/ median range to be provided.
Functional Assessment of Chronic Illness Therapy-General (FACT-G): Emotional | 3 months
  A 27-item self-related scale measure QoL across four domains of 'well-being' (physical, social/family, emotional and functional) on a 4-point Likert scale. Scores range from 0-24 for the emotional subscale. Data reported as continuous measure: means, standard deviation/ median range to be provided.
Mindfulness Attention Awareness Scale (MAAS) | 3 months
  A 15-item scale, designed to assess characteristics associated with mindfulness, such as: open or receptive awareness of and attention to what is taking place in the present. Participants use a scale from 1 to 6 (almost always - almost never), to indicate how frequently or infrequently they have each experience. Higher scores reflect higher levels of dispositional mindfulness. Data reported as continuous measure: means, standard deviation/ median range to be provided.
Brief Fatigue Inventory (BFI): Fatigue severity | 3 months
  This 9-item, 11-point rating scale was developed to assess subjective fatigue. The first three questions measure fatigue severity from 0, indicating "no fatigue," to 10, indicating "as bad as you can imagine," at current, usual, and worst levels. The following six questions assess fatigue interference with daily activities including general activity, mood, walking ability, normal work (both inside and outside the home), relations with other people, and enjoyment of life. Response options range from 0, indicating "does not interfere," to 10, indicating, "completely interferes." Higher scores on the BFI correspond to greater self-reported levels of fatigue. The time period for all questions is over the past 24 hours. Data reported as continuous measure: means, standard deviation/ median range to be provided.
Brief Fatigue Inventory (BFI): Fatigue Interferance | 3 months
  This 9-item, 11-point rating scale was developed to assess subjective fatigue. The first three questions measure fatigue severity from 0, indicating "no fatigue," to 10, indicating "as bad as you can imagine," at current, usual, and worst levels. The following six questions assess fatigue interference with daily activities including general activity, mood, walking ability, normal work (both inside and outside the home), relations with other people, and enjoyment of life. Response options range from 0, indicating "does not interfere," to 10, indicating, "completely interferes." Higher scores on the BFI correspond to greater self-reported levels of fatigue. The time period for all questions is over the past 24 hours. Data reported as continuous measure: means, standard deviation/ median range to be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta K Pal, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States